CLINICAL TRIAL: NCT04794673
Title: Cortex Motor Function Reorganization in Stroke Patients: A Longitudinal fMRI Study
Brief Title: Cortex Motor Function Reorganization in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Yan Liu, Department director, Guangzhou General Hospital of Guangzhou Military Command
Other Study IDs: LY-81825105
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2020-03

CONDITIONS: Ischemic Stroke
Keywords: motor cortex reorganization, Ischemic Stroke, fMRI, BOLD
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Left damage: Have the brain damage and the location of the damage in the left brain
  Interventions: Other: brain damage
- Right damage: Have the brain damage and the location of the damage in the right brain
  Interventions: Other: brain damage
- Nomal control: Not have the brain damage
  Interventions: Other: brain damage

INTERVENTIONS:
Other: brain damage — Have or not have the brain damage and the location of the damage

SUMMARY:
In China, stroke is among the highest morbidity and mortality, especially in senile population. Most of those patients had survived with various degrees of cerebral dysfunction; among them about 50% were motor deficit. Previous in vitro studies indicated that recovery of motor function after stroke were related not only to axonal regeneration or synapse reformation, but also functional reorganization of adjacent areas and other functional associated areas. The previous fMRI studies shown that the cerebral motor cortex possess the natural ability of self compensation and self reorganization in the situation of brain damage. It was characterized by equally bilateral activation in acute stage to partial ipsilateral activation and major contralateral activation in subacute stage to contralateral activation in chronic stage.

We plan to recruit first-episode acute cerebral infarction patients with single lesion on middle cerebral artery supply area and age and sex matched healthy volunteers. All the patients are going to assess in three different sessions (V1, 3 days after the onset of complaint, V2,30 days after onset of complaint; V3, 90 days after onset of the complaint ) with both clinical check as well as fMRI scan. The clinical assessment including dynamometer and finger tapping test to evaluate the strength and the flexibility of each upper legs and it also included the corresponding scales to exclude poststroke dementia and moderate and serious poststroke depression. The fMRI is scanned by using bilateral arm motor tasks. Motor cortex activation regions, activation of voxel between healthy controls and patients in different checkpoint are collected.

The purpose of this study is to investigate the dynamic process of motor cortical functional reorganization after cerebral stoke using functional magnetic resonance imaging combined with the behavior assessment. Meanwhile，we also studied the differences of motor function recovery and motor cortex compensation between dominant hemisphere and non-dominant hemisphere after stroke. Therefore, we could provide a theoretical basis and build up a useful evaluation system for rehabilitation after stroke and other arious cerebral injury.

DETAILED DESCRIPTION:
The cases derive from patients with acute ischemic stroke hospitalized in Neurology Department General Hospital of Guangzhou Military Command of PLA. The diagnosis of ischemic stroke is diagnosed using the diagnostic criteria of the International Association of Neurological Diseases and Stroke Association in 1982. The classification criteria for ischemic stroke are based on the current international TOAST etiological classification method.

The study passed the approval of the ethics committee of General Hospital of Guangzhou Military Command of PLA, and all patients or their guardian sign informed consent. According to the location and diagnostic criteria, the patients are divided into three groups: left hemisphere infarction patients group, right hemisphere infarction patients group and normal healthy control group. The subjects performed index finger tapping test, the maximum hand grip strength test of both hands, National Institute of Health stroke scale(NIHSS), Barthel Index(BI), Hamilton Anxiety Scale(HAMA), Hamilton Anxiety Scale(HAMA) and functional magnetic resonance (fMRI) tests at 3 days (V1), 30 days (V2) and 90 days (V3 phase) after the onset of cerebral infarction. In the healthy control group, the above examination is performed only 1 times. All subjects are assessed for clinical behavior by an independent third party.

Task-state function magnetic resonance design: Using the block design. There are two sequences. One sequence is in the way of rest and left hand movement, then repeat 5 times, ending at rest. The other is in the way of rest and right hand movement, then repeat 5 times, ending at rest. Each sequence lasted 220s, and the total duration of all tests was 440s. At the hand movement stage, each participant is at 1HZ Rhythm for the clenched fist movement with maximum strength, keep their whole body relaxed at the resting phase, with wrist and fingers not moving. participants use visual information to strictly control time and frequency of movement. Visual information is written by DMDX software, and accept the work instruction then sent to a transparent screen via a computer projector. Participants observed the information through a reflector mounted on a head coil.

Magnetic resonance data acquisition: 1.5 Tesla superconducting magnetic resonance scanner of Siemens Sonata company is applied. The standard phased array head coil is the radio frequency coil. Gradient field is 40m T/m, and switching rate is 200m T/m/ms. The scanning sequence and parameters are as follows:(1) T1 WI scan, obtaining whole brain structure image data: repeat time is 683ms, echo time is 11ms, layer thickness is 4mm, layer spacing is 1mm, matrix is 192x144, field of vision is 230mmx230mm, a total of 28 layers, range including whole brain. (2) The blood oxygen level dependent signal of the motor task state and resting state functional magnetic resonance imaging: using gradient echo combined with single excitation echo plane Imaging technology, the parameters are as follows: repeat time is 2000ms, echo time is 49ms, layer thickness is 4mm, layer spacing is 1mm, matrix is 64x64, field of vision is 210mmx210mm, a total of 28 layers.

ELIGIBILITY:
Inclusion Criteria:

* The first onset, the lesion was the single lesion of infarction or hemorrhage confirmed by head Magnetic Resonance Imaging(MRI) or Computed Tomography(CT).
* Hemiplegic hand muscle strength above grade 3, and was able to cooperate with the stimulation task of f MRI examination.
* According to the Edinburgh Handedness Questionnaire (EHQ) as the right hand.
* According to the commonly used eye chart examination, the naked eye vision >4.9.
* There is no central nervous system organic disease and other motor diseases that can affect hand function.
* No previous long-term alcoholism and long-term use of central nervous system activity and other drugs treatment.
* No contraindication to MRI scan.
* The patient cooperated with the examination and the patient or their guardian signed an informed consent.

Exclusion Criteria:

* Previous diseases of the central nervous system and peripheral nervous system that significantly affected the motor function of limbs.
* Significant cognitive impairment, MMSE≤27.
* Subjects was engaged in professional music playing or keyboard operation before illness.
* The level of consciousness drops after the illness.
* Significant anxiety and depression status (Hamilton anxiety scale ≥14 points, Hamilton depression scale ≥13 points) and other mental illness and history.
* Aphasia and neglect.
* History of epilepsy
* History of drug dependence
* Liver dysfunction, renal dysfunction, heart failure or other important organ function loss compensation
* Contraindication to MRI scan.
* Refuse to provide written consent or fail to cooperate with inspection for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to recruite first-episode acute cerebral infarction patients with single lesion on middle cerebral artery supply area and age and sex matched healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
A change of outcome measure: Index finger tapping test | This is an outcome measure to assess the improvement of motor function from onset to 3 months after treatment. Thus, participates will undergo this assessment on the 3 days (V1), 30 days (V2), and 90 days (V3) after randomization.
  The primary measure is the number of clicks that one index finger makes on the mouse as quickly as possible in 10 seconds.The subject took a sitting position and tapped the mouse with his index finger to record the fastest number of taps within 10 seconds.
A change of outcome measure: The maximum hand grip strength test | This is an outcome measure to assess the improvement of motor function from onset to 3 months after treatment. Thus, participates will undergo this assessment on the 3 days (V1), 30days (V2), and 90 days (V3) after randomization.
  Grip dynamometer(Beijing xintong sport equipment co. LTD, WCS-99.9 digital display electric the child dynamometer), in kilograms. To facilitate the maximum grip strength of one hand, the patient may place the arm in any position during the measurement, no body contact, elbows may be flexed or extended.

SECONDARY OUTCOMES:
A change of outcome measure: Functional Magnetic Resonance Imaging(fMRI) | We must determine that the participant is not in moderate or more cognitive impairment at each follow-up. Thus, participates will undergo this assessment on the 3 days (V1), 30 days (V2), and 90 days (V3) after randomization.
  The examine included task-state fMRI and resting-state fMRI Time Frame: We will explore the mechanisms of dynamic changes in language functions. Thus, participates will undergo this examine on the 3days (V1), 30 days (V2), and 90days (V3) after randomization.
National Institute of Health stroke scale(NIHSS ) | In order to ensure that participants can cooperate with our study, this assessment will be performed before randomization.
  The National Institutes of Health Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.NIHSS Scoring Instructions:0=No stroke symptoms, 1-4=Minor stroke, 5-15=Moderate stroke, 16-20=Moderate to severe stroke, 21-42=Severe stroke(i.e., The higher the score, the more severe the stroke).
Follow-up measurement: Hamilton Depression Rating Scale (HAMD) | We must determine that the participant is not in depression at each follow-up. Thus, participates will undergo this assessment on the 3 days (V1), 30 days (V2), and 90 days (V3) after randomization.
  The Hamilton Depression Rating Scale (HAMD) has proven useful for many years as a way of determining a patient's level of depression before, during, and after treatment. It generally takes 15-20 minutes to complete the interview and score the results. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine items are scored from 0-2. HAMD Scoring Instructions:0-7=Normal, 8-13 = Mild Depression, 14-18 = Moderate Depression, 19-22 = Severe Depression, ≥ 23 = Very Severe Depression(i.e.,the higher the score, the greater the likelihood of depression).
Follow-up measurement: Hamilton Anxiety Rating Scale (HAMA) | We must determine that the participant is not in anxiety at each follow-up. Thus, participates will undergo this assessment on the 3 days (V1), 30 days (V2), and 90 days (V3) after randomization.
  The Hamilton Anxiety Rating Scale (HAMA) is a widely used and well-validated tool for measuring the severity of a patient's anxiety. The HAMA is composed of 14 items and takes 15-20 minutes to complete the interview and score the results. Each item is scored on a 5-point scale, ranging from 0=not present to 4=severe.HAMA Scoring Instructions:0-8=Normal, 8-13= Possible Anxiety, 14-17 = Mild Anxiety, 18-24 = Moderate Anxiety, 25-30 = Severe Anxiety(i.e.,the higher the score, the greater the likelihood of anxiety).
Follow-up measurement: Mini-Mental State Examination (MMSE) | We must determine that the participant is not in moderate or more cognitive impairment at each follow-up. Thus, participates will undergo this assessment on the 3 days (V1), 30 days (V2), and 90 days (V3) after randomization.
  The Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. Administration of the test takes between 5 and 10 minutes. The MMSE test includes simple questions and problems in a number of areas: the time and place of the test, repeating lists of words, arithmetic such as the serial sevens, language use and comprehension, and basic motor skills. Any score greater than or equal to 24 points (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.The raw score may also need to be corrected for educational attainment and age.

CONTACTS AND LOCATIONS:
Overall Officials: Yan LIU, PhD, Study Chair — Guangzhou General of Guangzhou Military Command
Locations (1):
- General Hospital of Southern Theatre Command,PLA, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brown DL, Lisabeth LD, Garcia NM, Smith MA, Morgenstern LB. Emergency department evaluation of ischemic stroke and TIA: the BASIC Project. Neurology. 2004 Dec 28;63(12):2250-4. doi: 10.1212/01.wnl.0000147292.64051.9b. PMID 15623682
- [Background] Kokotilo KJ, Eng JJ, McKeown MJ, Boyd LA. Greater activation of secondary motor areas is related to less arm use after stroke. Neurorehabil Neural Repair. 2010 Jan;24(1):78-87. doi: 10.1177/1545968309345269. Epub 2009 Sep 8. PMID 19737873
- [Background] Swayne OB, Rothwell JC, Ward NS, Greenwood RJ. Stages of motor output reorganization after hemispheric stroke suggested by longitudinal studies of cortical physiology. Cereb Cortex. 2008 Aug;18(8):1909-22. doi: 10.1093/cercor/bhm218. Epub 2008 Jan 29. PMID 18234688
- [Background] O'Shea J, Johansen-Berg H, Trief D, Gobel S, Rushworth MF. Functionally specific reorganization in human premotor cortex. Neuron. 2007 May 3;54(3):479-90. doi: 10.1016/j.neuron.2007.04.021. PMID 17481399
- [Background] Lotze M, Markert J, Sauseng P, Hoppe J, Plewnia C, Gerloff C. The role of multiple contralesional motor areas for complex hand movements after internal capsular lesion. J Neurosci. 2006 May 31;26(22):6096-102. doi: 10.1523/JNEUROSCI.4564-05.2006. PMID 16738254
- [Background] Cramer SC, Nelles G, Benson RR, Kaplan JD, Parker RA, Kwong KK, Kennedy DN, Finklestein SP, Rosen BR. A functional MRI study of subjects recovered from hemiparetic stroke. Stroke. 1997 Dec;28(12):2518-27. doi: 10.1161/01.str.28.12.2518. PMID 9412643
- [Background] Rossini PM, Dal Forno G. Integrated technology for evaluation of brain function and neural plasticity. Phys Med Rehabil Clin N Am. 2004 Feb;15(1):263-306. doi: 10.1016/s1047-9651(03)00124-4. PMID 15029909
- [Background] Nelles G, Spiekramann G, Jueptner M, Leonhardt G, Muller S, Gerhard H, Diener HC. Evolution of functional reorganization in hemiplegic stroke: a serial positron emission tomographic activation study. Ann Neurol. 1999 Dec;46(6):901-9. doi: 10.1002/1531-8249(199912)46:63.0.co;2-7. PMID 10589543
- [Background] Calautti C, Leroy F, Guincestre JY, Baron JC. Dynamics of motor network overactivation after striatocapsular stroke: a longitudinal PET study using a fixed-performance paradigm. Stroke. 2001 Nov;32(11):2534-42. doi: 10.1161/hs1101.097401. PMID 11692013
- [Background] Marshall RS, Perera GM, Lazar RM, Krakauer JW, Constantine RC, DeLaPaz RL. Evolution of cortical activation during recovery from corticospinal tract infarction. Stroke. 2000 Mar;31(3):656-61. doi: 10.1161/01.str.31.3.656. PMID 10700500
- [Background] Taub E, Miller NE, Novack TA, Cook EW 3rd, Fleming WC, Nepomuceno CS, Connell JS, Crago JE. Technique to improve chronic motor deficit after stroke. Arch Phys Med Rehabil. 1993 Apr;74(4):347-54. PMID 8466415
- [Background] Liepert J, Bauder H, Wolfgang HR, Miltner WH, Taub E, Weiller C. Treatment-induced cortical reorganization after stroke in humans. Stroke. 2000 Jun;31(6):1210-6. doi: 10.1161/01.str.31.6.1210. PMID 10835434
- [Background] Rouiller EM, Yu XH, Moret V, Tempini A, Wiesendanger M, Liang F. Dexterity in adult monkeys following early lesion of the motor cortical hand area: the role of cortex adjacent to the lesion. Eur J Neurosci. 1998 Feb;10(2):729-40. doi: 10.1046/j.1460-9568.1998.00075.x. PMID 9749734
- [Background] Nudo RJ, Milliken GW. Reorganization of movement representations in primary motor cortex following focal ischemic infarcts in adult squirrel monkeys. J Neurophysiol. 1996 May;75(5):2144-9. doi: 10.1152/jn.1996.75.5.2144. PMID 8734610
- [Background] Brasil-Neto JP, Valls-Sole J, Pascual-Leone A, Cammarota A, Amassian VE, Cracco R, Maccabee P, Cracco J, Hallett M, Cohen LG. Rapid modulation of human cortical motor outputs following ischaemic nerve block. Brain. 1993 Jun;116 ( Pt 3):511-25. doi: 10.1093/brain/116.3.511. PMID 8513390
- [Background] Nelles G, Jentzen W, Jueptner M, Muller S, Diener HC. Arm training induced brain plasticity in stroke studied with serial positron emission tomography. Neuroimage. 2001 Jun;13(6 Pt 1):1146-54. doi: 10.1006/nimg.2001.0757. PMID 11352620
- [Background] Karni A, Meyer G, Jezzard P, Adams MM, Turner R, Ungerleider LG. Functional MRI evidence for adult motor cortex plasticity during motor skill learning. Nature. 1995 Sep 14;377(6545):155-8. doi: 10.1038/377155a0. PMID 7675082
- [Background] Johansen-Berg H, Dawes H, Guy C, Smith SM, Wade DT, Matthews PM. Correlation between motor improvements and altered fMRI activity after rehabilitative therapy. Brain. 2002 Dec;125(Pt 12):2731-42. doi: 10.1093/brain/awf282. PMID 12429600
- [Background] Enzinger C, Dawes H, Johansen-Berg H, Wade D, Bogdanovic M, Collett J, Guy C, Kischka U, Ropele S, Fazekas F, Matthews PM. Brain activity changes associated with treadmill training after stroke. Stroke. 2009 Jul;40(7):2460-7. doi: 10.1161/STROKEAHA.109.550053. Epub 2009 May 21. PMID 19461018
- [Background] James GA, Lu ZL, VanMeter JW, Sathian K, Hu XP, Butler AJ. Changes in resting state effective connectivity in the motor network following rehabilitation of upper extremity poststroke paresis. Top Stroke Rehabil. 2009 Jul-Aug;16(4):270-81. doi: 10.1310/tsr1604-270. PMID 19740732
- [Background] Page SJ, Harnish SM, Lamy M, Eliassen JC, Szaflarski JP. Affected arm use and cortical change in stroke patients exhibiting minimal hand movement. Neurorehabil Neural Repair. 2010 Feb;24(2):195-203. doi: 10.1177/1545968309360501. PMID 20107135
- [Background] Page SJ, Szaflarski JP, Eliassen JC, Pan H, Cramer SC. Cortical plasticity following motor skill learning during mental practice in stroke. Neurorehabil Neural Repair. 2009 May;23(4):382-8. doi: 10.1177/1545968308326427. Epub 2009 Jan 20. PMID 19155350
- [Background] Michielsen ME, Selles RW, van der Geest JN, Eckhardt M, Yavuzer G, Stam HJ, Smits M, Ribbers GM, Bussmann JB. Motor recovery and cortical reorganization after mirror therapy in chronic stroke patients: a phase II randomized controlled trial. Neurorehabil Neural Repair. 2011 Mar-Apr;25(3):223-33. doi: 10.1177/1545968310385127. Epub 2010 Nov 4. PMID 21051765
- [Background] Mattson MP, Maudsley S, Martin B. BDNF and 5-HT: a dynamic duo in age-related neuronal plasticity and neurodegenerative disorders. Trends Neurosci. 2004 Oct;27(10):589-94. doi: 10.1016/j.tins.2004.08.001. PMID 15374669
- [Background] Goldstein LB. Effects of amphetamines and small related molecules on recovery after stroke in animals and man. Neuropharmacology. 2000 Mar 3;39(5):852-9. doi: 10.1016/s0028-3908(99)00249-x. PMID 10699450
- [Background] Coppell AL, Pei Q, Zetterstrom TS. Bi-phasic change in BDNF gene expression following antidepressant drug treatment. Neuropharmacology. 2003 Jun;44(7):903-10. doi: 10.1016/s0028-3908(03)00077-7. PMID 12726822
- [Background] Semkova I, Wolz P, Krieglstein J. Neuroprotective effect of 5-HT1A receptor agonist, Bay X 3702, demonstrated in vitro and in vivo. Eur J Pharmacol. 1998 Oct 23;359(2-3):251-60. doi: 10.1016/s0014-2999(98)00634-7. PMID 9832397
- [Background] Cheng YD, Al-Khoury L, Zivin JA. Neuroprotection for ischemic stroke: two decades of success and failure. NeuroRx. 2004 Jan;1(1):36-45. doi: 10.1602/neurorx.1.1.36. PMID 15717006
- [Background] Chang YC, Tzeng SF, Yu L, Huang AM, Lee HT, Huang CC, Ho CJ. Early-life fluoxetine exposure reduced functional deficits after hypoxic-ischemia brain injury in rat pups. Neurobiol Dis. 2006 Oct;24(1):101-13. doi: 10.1016/j.nbd.2006.06.001. Epub 2006 Aug 2. PMID 16887358
- [Background] Boyeson MG. Effects of fluoxetine and maprotiline on functional recovery in poststroke hemiplegic patients undergoing rehabilitation therapy. Stroke. 1996 Nov;27(11):2145-6. No abstract available. PMID 8898832
- [Background] Pariente J, Loubinoux I, Carel C, Albucher JF, Leger A, Manelfe C, Rascol O, Chollet F. Fluoxetine modulates motor performance and cerebral activation of patients recovering from stroke. Ann Neurol. 2001 Dec;50(6):718-29. doi: 10.1002/ana.1257. PMID 11761469